CLINICAL TRIAL: NCT05959369
Title: Investigation of Relationship Between Balance, Core Stabilization and Foot Posture in Kickboxers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, KÜBRA USLU, physiotherapist, Uskudar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 61351342/MART 2023-27
Record Dates: First submitted 2023-06-13; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: description study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elite kickboxer (Experimental): athletes who have completed the age of 18 professionally, participating in fighting competitions and actively training
  Interventions: Diagnostic Test: y balance test, core endurance and strength test, foot posture ındex

INTERVENTIONS:
Diagnostic Test: y balance test, core endurance and strength test, foot posture ındex — First, the athlete's bare feet will be photographed on a flat surface for foot posture analysis. Modified push-up test and sit-up test will be used for core stabilization evaluation. For the endurance assessment of core muscles, lateral bridge test, static trunk extension test (Sorensen test) and trunk flexors endurance test will be used. The 'Y' balance test will be used for balance evaluation. The athlete will be asked to lie in three different directions at the same time with the other foot while balancing on one foot.

SUMMARY:
This study aimed to investigate relationship between balance, core stabilization and foot posture in kickboxers. This descriptive study was planned to be conducted to 40 elite athletes as volunteer.

DETAILED DESCRIPTION:
Based on self-defense with weighted kicks and punches, developed by breathing from kickboxing, karate, thai boxing and western boxing; balance, condition and agility requirements are one of the modern combat sports. Athletes who practice at high exercise intensity need strong motor skills, a developed aerobic and anaerobic physical capacity, and excellent tactile senses. A typical kickboxing tournament consists of 3-12 rounds lasting 2-4 minutes with 1 rest period between rounds. In standing combat sports, body posture represents a certain harmony of lower and upper body positions. These contact sports injuries have a very high risk of injury. ). In a study conducted by Lystad in 2015 on kickboxers, it was reported that the overall injury incidence was 39% and the most frequently injured anatomical regions were the head (57.8%) and lower extremities (26.1%).

The core system muscles are a system that provides the power between the lower and upper half of the trunk, provides body stability, and forms all other muscle structures of 29 different muscles. Local stabilization and global stabilization are divided into system muscles. local stabilization muscles; M. Transverse abdominis, m. Internal oblique, m. Multifidus can be taken from and from the pelvic floor muscles. Global stabilization muscles; quadratus lumborum, internal and external oblique, gluteus medius and adductor muscles. Core stabilization muscles assist spinal stability by increasing abdominal pressure and weights in the thoracolumbar fascia, supporting spinal stability finals, spinal intersegment falling forces and excessive pressure endings. The speed with which the core muscles provide stability to the body has a direct bearing on the strength and coordination of extreme movement. However, in the literature, the parts where core stabilization muscles are not missing are at the point where lower extremity injuries occur more.

The balance may be termed the shield to hold the body center of gravity within the stability frames drawn by the support base. It is known that balance, which is an important parameter in the realization of daily life behaviors, plays an important role in the emergence of postural control, changing direction, moving the object, and many sports skills and advanced movements. To control balance, the central nervous system contributes to balance control, which can combine visual, vestibular and proprioceptive information to elicit motor commands that govern the movement of muscles. Thus, it plays an important role in balance control by determining the position of the hand and movements in space. Theoretically, the body is located everywhere proprioceptive information distribution to balance control.

Enhanced core stabilization and balance allow for maximum force output, increased neuromuscular efficiency, the benefits of their overhead, efficient biomechanical function, and the consequences of their overuse. It also provides more efficient, accurate and powerful movements by limiting the use of the upper and lower extremity muscles of the athletes.

Mcgill once again argued that lumbar injuries can be reduced by improving the stability and coordination of the deep abdominal muscles that are effective in protecting and maintaining core stabilization injuries.

Foot type affects lower extremity functions, groups and functional smoothness, and the entire biomechanical chain of the body. Foot and ankle injuries can cause deterioration of balance and body posture. The heart foot cells in the clinic center are anatomically divided into three groups as foot supination, foot pronation and neutral foot. During most sports regulation, the foot is the only part of the mechanical body that touches the ground, and the complex motor processors required in elite sports receive the necessary information to enable upper body movements in addition to foot positions to be successful. The deterioration of the foot appearance affects and changes the foot structure of its long time.

As a result, it has been determined that poor balance ability is a factor associated with an increased risk of foot complex injury. In another study, it was concluded that individuals with foot supination or pronation had lower static postural control on one foot compared to individuals with neutral feet, and it was emphasized that these muscles should be given special importance in the rehabilitation of lower extremity injuries. Mulligan et al. (2013) and Hashimoto et al. (2014) conducted studies showing that by strengthening the intrinsic and extrinsic muscles of the foot, the height and shape of the MLA will be positively affected, and balance and performance will increase.

In martial arts, long-term training load can lead to sport-specific functional and body posture adaptations. The importance of evidence-based information about these functional and body posture adaptations comes to the fore in the rehabilitation and treatment process. Despite its popularity, there is a paucity of published data describing kickboxing injury patterns and the etiology of injuries.

Although there are limited studies examining balance and core stabilization in kickboxers, there is no study evaluating the relationship between foot posture, core stabilization and balance with foot posture.

ELIGIBILITY:
Inclusion Criteria:

* professionale kickboxers

Exclusion Criteria:

* unadult

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-18 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
test scores | 1 year
  relationship between core stabilization scores (repetitions in 30 seconds) and y balance test scores ( centimeters)

IPD SHARING:
Plan to Share IPD: No
no sharing